CLINICAL TRIAL: NCT02247141
Title: A Multi-centre Open Study to Assess the Safety and Efficacy of Subgam® Given Via the Subcutaneous Route in Primary Antibody Deficient Patients.
Brief Title: A Multi-centre Open Study to Assess the Safety and Efficacy of Subgam®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: SCIG01
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Primary Antibody Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

ARMS (1):
- Subgam® (Experimental)
  Interventions: Biological: Subgam® (Human Normal Immunoglobulin Solution)

INTERVENTIONS:
Biological: Subgam® (Human Normal Immunoglobulin Solution)

SUMMARY:
The primary objective was to determine the efficacy of Human Normal Immunoglobulin (Subgam®) given subcutaneously by weekly infusion to patients with primary antibody deficiency.

The secondary objective was to determine the safety of Subgam® given subcutaneously by weekly infusion to patients with primary antibody deficiency.

ELIGIBILITY:
Inclusion Criteria:

* The main criteria for inclusion in the study were as follows:

  * A diagnosis of primary antibody deficiency;
  * No lower or upper age limit (any age was eligible);
  * With stable disease and receiving immunoglobulin (IVIG or SCIG) therapy for at least six months prior to starting the study;
  * Written informed consent (patient/parent/guardian).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Proportion of trough levels at each time point where serum IgG was more than equal to 4 g/L | Before each infusion in the first 6 months of the study (approximately 30 infusions)

CONTACTS AND LOCATIONS:
Locations (14):
- United Kingdom (14):
  - Papworth Hospital, Papworth Everard, Cambridgeshire
  - Royal Preston Hospital, Preston, Lancashire
  - Guest Hospital, Dudley, West Midlands
  - Birmingham Children's Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - St James' University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Great Ormond Street Hospital, London
  - St Bartholomew's Hospital, London
  - John Radcliffe Hospital, Oxford
  - Hope Hospital, Salford
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - St Helier Hospital, Carshalton, Surrey

REFERENCES:
- [Derived] Dash C, Gascoigne E, Gillanders K, Gooi H. Experience with Subgam, a Subcutaneously Administered Human Normal Immunoglobulin (ClinicalTrials.gov--NCT02247141). PLoS One. 2015 Jul 29;10(7):e0131565. doi: 10.1371/journal.pone.0131565. eCollection 2015. PMID 26222441
- See also: Related Info — http://www.bpl.co.uk